CLINICAL TRIAL: NCT05654922
Title: A Phase 3, Open-label, Randomized, Standard of Care-controlled, Parallel Study Arm Study to Demonstrate Efficacy and Safety of ARINA-1 in the Prevention of Bronchiolitis Obliterans Syndrome (BOS) Progression in Participants With a Bilateral Lung Transplant
Brief Title: Study to Evaluate ARINA-1 in the Prevention of Bronchiolitis Obliterans Progression in Participants With Bilateral Lung Transplant
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Renovion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RVN-001
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Pre-Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: For individuals performing spirometry, every attempt will be made to keep them masked to treatment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARINA-1 plus standard of care (Experimental): ARINA-1 (88 mg/mL ascorbic acid, ASC; 150 mg/mL reduced glutathione, GSH); fixed dose, 4 mL solution inhaled twice daily via nebulization plus standard 3-therapy immunosuppression regimen and azithromycin
  Interventions: Drug: ARINA-1
- Standard of care only (Other): Standard 3-therapy immunosuppression regimen and azithromycin
  Interventions: Other: Standard of care only

INTERVENTIONS:
Drug: ARINA-1 — ARINA-1 (88 mg/mL ascorbic acid, ASC; 150 mg/mL reduced glutathione, GSH)
  Arms: ARINA-1 plus standard of care
Other: Standard of care only — Standard 3-therapy immunosuppression regimen and azithromycin
  Arms: Standard of care only

SUMMARY:
The goal of this Phase 3 clinical trial is to compare ARINA-1 (a nebulized immunomodulatory agent) plus Standard of Care vs Standard of Care alone. The main question it aims to answer are:

* Evaluate the effectiveness of ARINA-1 in preventing bronchiolitis obliterans syndrome (BOS) progression in participants with a bilateral lung transplant
* To evaluate the effectiveness of ARINA-1 on improving quality of life decline and preventing or delaying the use of augmented immunosuppression in participants with pre-BOS relative to SOC.

Participants will have clinic visits at screening, randomization (day 1) and weeks 4, 12, 18, and 24. After week 24, participants will have clinic visits at weeks 32, 40, and 48.

Participants will also have a telehealth visit on day 2 and phone calls to assess adverse events (AEs), serious adverse events (SAEs), and review patient education will occur during weeks 5, 8, 36, and 44.

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral lung transplant >12 months from the time of Visit 1 / Randomization
2. Age 18-75 years old at the time of consent
3. Routinely followed at enrolling site
4. Willing and able to comply with visit schedule and at-home requirements
5. 10-24% decrease in FEV1 from the post-transplant baseline within the last 12 months.
6. Capable of giving informed consent
7. On a stable maintenance regimen of azithromycin for >4 weeks prior to the Screening Visit
8. On a stable 2-agent or 3-agent immunosuppression regimen that includes a steroid, a calcineurin inhibitor (CNI), and, optionally, a cell cycle inhibitor (e.g., mycophenolate, azathioprine) >4 weeks prior to Screening
9. If a woman of childbearing potential (WOCBP), must agree to use a reliable method of birth control for the entire duration of the study.

Exclusion Criteria:

1. Positive urine pregnancy test at screening and baseline visit
2. Diagnosis of active congestive heart failure or symptomatic coronary artery disease > grade 3 based on the New York Heart Association Functional Classification (NYHA) criteria
3. Restrictive allograft syndrome (RAS) defined by radiographic interstitial or alveolar opacities on chest X-ray or CT scan that are consistent with RAS
4. Have advanced BOS, defined by >24% decrease in FEV1 in post-transplant baseline
5. A diagnosis of probable antibody-mediated rejection (AMR) <12 months prior to the baseline visit
6. Donor-specific antibodies (DSA) identified <6 months prior to the baseline visit. *The presence of DSA >6 months from the baseline visit is acceptable for enrollment into the study.
7. Unresolved diffuse alveolar damage
8. Receiving mechanical ventilation
9. Chronic kidney disease stage IV or higher, including on dialysis
10. Initiating a new maintenance therapy or changing immunosuppression maintenance therapy (e.g., changing tacrolimus to cyclosporine) <30 days prior to the baseline visit.
11. Have initiated or changed mTOR maintenance therapy <3 months prior to Clinic Visit 1 (mTOR use for >3 months is allowed)
12. Initiating or changing antibiotic (including azithromycin), antiviral, or antifungal therapy <14 days prior to the baseline visit.
13. Use of alemtuzumab <6 months prior to the baseline visit
14. Use of anti-thymocyte therapies (e.g., anti-thymocyte globulin) or photopheresis <90 days prior to the Screening Visit. Prior use of Trikafta (elexacaftor, ivacaftor, and tezacaftor is allowed as long as the participant has been on stable dose for >90 days prior to the Screening Visit.
15. Initiating a multivitamin or other supplement (inhaled, oral, or IV) containing vitamin C, glutathione, or N-acetylcysteine <90 days prior to the baseline visit
16. Significant unstable comorbidities, in the opinion of the site investigator
17. Allery or previous adverse reaction to azithromycin
18. A diagnosis of dynamic collapse / tracheobrochomalacia <90 days of the baseline visit.
19. Subjects currently participating in, or who have participated in an interventional (drug or device) clinical study <30 days of the baseline visit.
20. Have been diagnosed with ARAD within 6 weeks of the Screening Visit.
21. Have used belatacept <6 months prior to Clinic Visit 1
22. Have had an initial treatment of bronchial stents or cryotherapy within 12 months of the Screening Visit, or had bronchial stents removed within the last 3 months of the Screening Visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Percentage change from baseline in FEV1 (%ΔFEV1) | 24 weeks
  Week 24 (mL) - Baseline (mL) = ΔFEV1 (mL) ΔFEV1 (mL) / Baseline (mL) x 100 = %ΔFEV1

SECONDARY OUTCOMES:
Percentage change from baseline of Forced Expiratory Volume in one second (FEV1) | 48 weeks
  Week 48 (mL) - Baseline (mL) = ΔFEV1 (mL) ΔFEV1 (mL) / Baseline (mL) x 100 = %ΔFEV1
Percentage change from baseline of Forced Vital Capacity (FVC) | 24 weeks
Percentage change from baseline of FVC | 48 weeks
Percentage change from baseline of FEF25-75% | 24 weeks
Percentage change from baseline of FEF25-75% | 48 weeks
Number of participants in each arm with augmented immunosuppression | 24 weeks
  number
Number of participants in each arm with augmented immunosuppression | 48 weeks
Time to initiation of augmented immunosuppression | over the duration of the 48 week trial
  Length of time to when participant requires a change in their immunosuppression regimen
Change from baseline in Saint George's Respiratory Questionnaire total score | 24 weeks
  quality of life questionnaire, total score of 0 to 100, higher score = more limitations
Change from baseline in Saint George's Respiratory Questionnaire total score | 48 weeks
  quality of life questionnaire, total score of 0 to 100, higher score = more limitations
Proportion of participants requiring the use of antimicrobial agents to treat a pulmonary infection | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tim Whelan, MD, Principal Investigator — Medical University of South Carolina
Locations (20):
- United States (20):
  - Dignity Health - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of California Los Angeles School of Medicine, Los Angeles, California
  - University of California San Diego Health, San Diego, California
  - Advent Health, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Hospital, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor Scott and White Research Institute, Dallas, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia